CLINICAL TRIAL: NCT01386541
Title: Investigation of Safety/Tolerability, Pharmacokinetics and Pharmacodynamics After Multiple Ascending Doses of BYK324677 in Healthy Volunteers. A Monocentre, Placebo-controlled, Cross-over, Double-blind, Randomised Trial
Brief Title: Multiple Ascending Dose Trial of BYK324677 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B5-8012-101-RD; 2010-023857-12 (EudraCT Number)
Record Dates: First submitted 2011-06-28; First posted 2011-07-01 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BYK324677 (Active Comparator): * Dose group I: total daily dose 2 mg (1 mg BID or 2 mg SID)
  * Dose group II: total daily dose 4 mg (2 mg BID or 4 mg SID)
  * Dose group III: total daily dose 6 mg (3 mg BID or 6 mg SID)
  In each dose group 12 subjects (8 subjects BYK324677, 4 subjects placebo) are planned.
  Within each dose group, the subjects will be randomised to either BYK324677 or placebo at a ratio of 2:1.
  Within each verum group, the subjects will be randomised to one of the 2 treatment sequences (BID/SID or SID/BID, ratio 1:1) and treated in a cross-over manner.
  Interventions: Drug: BYK324677
- Placebo (Placebo Comparator)
  Interventions: Drug: BYK324677

INTERVENTIONS:
Drug: BYK324677 — capsules, administered orally

SUMMARY:
This monocenter trial is conducted to obtain first data on safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) after multiple ascending doses of BYK324677 in humans. In addition, the trial should provide preliminary information on a possible influence of sex, food intake, and posology (once or twice daily administration of BYK324677) to support the further planning of the drug development programme.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent
* Healthy male and female subjects. Assessed as healthy based on a screening examination including medical history, physical examination, blood pressure (systolic ≤140 mmHg, diastolic ≤90 mmHg), pulse rate (within 45-95 bpm), ECG assessment, and clinical laboratory results
* Body mass index (BMI) between ≥18 and ≤28 kg/m², and a body weight ≥60 kg

Exclusion Criteria:

* History or current evidence of specified diseases
* History of malignancy in the past 5 years
* Gain or loss in body weight of more than 5% within the last 2 months or use of weight-loss medication within the last 3 months
* ECG abnormalities of clinical relevance
* Suspected hypersensitivity to the trial medication
* Positive virology tests indicating acute or chronic infections
* Clinically relevant laboratory parameters outside a specified range
* Use of specified medications within certain time frames or use of certain co-medications
* Abuse of alcohol or drugs
* Dietary habits that would prevent from taking standardised meals
* Female subjects: positive pregnancy test; lack of medically reliable methods of contraception during the trial
* Donation of blood
* Smoking within the last 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety/tolerability of multiple dosing of BYK324677 given once daily (SID) or twice daily (BID) in healthy volunteers. | during screening, clinical part (treatment) and end-of-trial examination (up to 8 weeks)
  Safety/tolerability variables: adverse events (AEs), vital signs (BP, pulse rate, body temperature), 12-lead ECG (PQ [=PR], QRS, QT, QTcF and QTcB intervals, heart rate), laboratory parameters including urinalysis.

SECONDARY OUTCOMES:
Exploratory assessment of the pharmacokinetics (PK) of multiple dosing of BYK324677 (SID or BID) under steady state conditions in healthy volunteers. | during Treatment Period 1 and Period 2 (up to 3 weeks)
  Pharmacokinetic variables (e.g. AUC, Cmax, tmax, t1/2) of BYK324677 on Day 1 and Day 5 (single dose i.e. after first Investigational medicinal product (IMP) dose vs steady state) as well as on Day 4 and Day 5 (fed vs fasted, respectively).
Exploratory assessment of the pharmacodynamics (PD) of multiple dosing of BYK324677 (SID or BID) under steady state conditions in healthy volunteers. | during Treatment Period 1 and Period 2 (up to 3 weeks)
  Pharmacodynamic variables glucose, insulin, glucagon-like peptide 1 and glucagon on Day -1, Day 4 (fed) and Day 5 (fasted).

CONTACTS AND LOCATIONS:
Locations (1):
- Nycomed Investigational site, Mannheim, Germany